CLINICAL TRIAL: NCT02900222
Title: Study of Endoscopic Choroid Plexus Cauterization for Adult Patients With Hydrocephalus and Risk Factors for Perioperative Complications Following Shunt Surgery.
Brief Title: Study of Choroid Plexus Cauterization in Patients With Hydrocephalus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Resources no longer available
Sponsor: Ronald Benveniste (Other)
Responsible Party: Sponsor-Investigator, Ronald Benveniste, Associate Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20160650
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Choroid Plexus Coagulation (Experimental): Patients with communicating hydrocephalus will be treated with endoscopic choroid plexus coagulation.
  Interventions: Procedure: endoscopic choroid plexus coagulation

INTERVENTIONS:
Procedure: endoscopic choroid plexus coagulation — A burr hole will be made over the frontal lobe of the brain. An endoscope will be introduced into the ventricle of the brain and the choroid plexus coagulated with an electrocautery device. The septum pellucidum separating the right and left lateral ventricles will be opened, and the choroid plexus on the opposite side coagulated as well.

SUMMARY:
The purpose of this study is to determine whether endoscopic choroid plexus coagulation is safe in adult patients with communicating hydrocephalus and risk factors for complications from the standard surgical treatment. It may also help determine whether the endoscopic choroid plexus coagulation is effective in treating your communicating hydrocephalus. The Investigators hope that this research will allow us to place fewer shunts in patients with conditions similar to yours, avoiding complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 or older) with communicating hydrocephalus, who have risk factors for complications following shunt surgery. Risk factors include loculated hydrocephalus (i.e., imaging evidence that the ventricles of the brain do not communicate with each other, in the setting of known communicating hydrocephalus); prior episodes of ventriculitis and/or shunt infection; subdural hematoma associated with shunt placement; inability to place a distal catheter in the peritoneal cavity due to scarring or prior infection; and multiple prior episodes of shunt failure.
* In patients with communicating hydrocephalus who have significantly increased lateral and third ventricular size and normal fourth ventricular size, an endoscopic third ventriculostomy will be performed in conjunction with the choroid plexus cauterization, provided that communicating hydrocephalus is thought to be present, based on either the history (for example, past meningitis or other infectious or inflammatory disease, or history of communicating hydrocephalus without disproportion of the ventricles in the past; or imaging findings, such as patency of the foramina of Magendie and Luschka).

Exclusion Criteria:

* Exclusion criteria include patients who have non-communicating hydrocephalus; patients who are undergoing emergency surgery because of rapid decline in neurologic condition; and patients with medical conditions such as coagulopathy or severe cardiac conditions, that preclude neurosurgical intervention.
* In the case of adults unable to consent, informed consent will be obtained from appointed health care proxies. Minors, pregnant women, and prisoners will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Occurrence of post-operative complications | 30 days
  Complications will be defined as new neurologic deficits after surgery; hemorrhage or stroke on postoperative imaging studies; or other perioperative complications.

SECONDARY OUTCOMES:
Shunt independence | 1 year
  Shunt independence is defined as the patient surviving with no need for ventricular shunt placement

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Benveniste, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No